CLINICAL TRIAL: NCT03990376
Title: Establishment of a Gold Standard Formula for Blood Loss Calculation in Adolescent Idiopathic Scoliosis (AIS) Surgery
Brief Title: Adolescent Idiopathic Scoliosis (AIS) Gold Standard for Blood Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Nicholas Fletcher, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00101023
Record Dates: First submitted 2019-06-11; First posted 2019-06-19 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Scoliosis; Pediatric surgery; Orthopedics; Blood loss
MeSH Terms: conditions — Scoliosis; Hemorrhage

STUDY DESIGN:
Intervention Model Description: Participants include 45 adolescent subjects undergoing spinal fusion for correction of idiopathic scoliosis.
  After obtaining a baseline sample of 5 mL of blood, 1 mL of I-131-labeled albumin will be injected intravenously over 1 min. At the time the baseline sample is obtained, a hematocrit will be simultaneously acquired. Five milliliter blood samples will then be collected at 12, 18, 24, 30, and 36 min post-injection, and the Plasma volume (PV) will be measured by extrapolating to time zero. This entire process will occur twice per patient: once pre-procedure and once post-procedure.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Blood volume assessment with Blood Volume Analyzer (Other): Injections of 1 mL of I-131-labeled serum albumin based on each patient's height and weight - 1 pre-surgical and 1 post-surgical
  Interventions: Other: Radioisotope I-131-labeled albumin

INTERVENTIONS:
Other: Radioisotope I-131-labeled albumin — 1 mL of radioisotope I-131-labeled albumin x 2

SUMMARY:
The purpose of this study is to establish a benchmark for measuring blood loss by directly measuring the change in red cell volume before and after surgery and to compare established blood loss estimators to this benchmark in order to determine the most accurate and precise method for estimating blood loss in adolescent idiopathic scoliosis surgery patients

DETAILED DESCRIPTION:
Bleeding is a necessary and unavoidable part of spine surgery. It is important to the surgeons and anesthesiologists to know how much blood a patient has lost during surgery in order to care for them in the best way possible. Different methodology has been employed to estimate how much blood is lost during surgery, but unfortunately none of the methods used have been reliable. The study will calculate surgical blood loss by determining perioperative change in red cell volume that is directly measured by using a special method that relies on radioisotope I-131-labeled albumin administration (BVA-100) during the surgery. This benchmarked blood loss estimate will then be compared to estimates calculated using the Gross equation, the Bourke and Smith equation, and the Camarasa formula. In addition, blood loss will be estimated volumetrically by utilizing formulas based on the amount of salvaged blood produced by an intraoperative salvaging system (Cell Saver®). Blood loss estimates based on salvaged blood volume will also be compared to the benchmark.

ELIGIBILITY:
Inclusion Criteria:

* Ages 10-17 years old
* Surgery scheduled for posterior spinal fusion correction of idiopathic scoliosis

Exclusion Criteria:

* Congenital or neuromuscular scoliosis
* Known coagulopathy or platelet dysfunction

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
The change in blood loss (in mLs) determined by the benchmark technique (directly measured red cell volume loss by BVA-100 Blood Volume Analyzer divided by average intraoperative hematocrit) and each of an established set of blood loss estimators | Blood loss will be assessed immediately after surgery (closing of incision)
  The established blood loss estimators include the Gross equation, the Bourke and Smith equation, the Camarasa formula, and equations based on salvaged blood volumes (e.g. 2x cell saver volume). The benchmark blood loss estimate and all of the established blood loss estimators will estimate blood loss in mLs. Thus, the change in surgical blood loss between the benchmark estimator and each of the established blood loss estimators will also be in mLs.

SECONDARY OUTCOMES:
The change in pre-surgical blood volume (in mLs) directly measured by the BVA-100 Blood Volume Analyzer and each of an established set of blood volume estimators | Blood volume will be measured at the beginning of surgery (immediately after anesthetic induction)
  The established blood volume estimators include Moore's formula, Nadler's formula, and the International Council for Standardization in Haematology (ICSH) equation. The BVA-100 blood volume estimate and all of the established blood volume estimators will estimate blood volume in mLs. Thus, the change in preoperative blood volume between the BVA-100 estimate and each of the established blood volume estimators will also be in mLs.

OTHER OUTCOMES:
The ratio of red blood cell volume recovered by an intraoperative blood salvaging system (Cell Saver®) and the red cell volume lost (determined by BVA-100 Blood Volume Analyzer) during the surgery | Immediately after surgery (closing of incision)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Fletcher, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta - Egleston Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No